CLINICAL TRIAL: NCT05446532
Title: Characteristics of Hepatitis B HBsAg & HBsAc Carriers Simultaneously
Brief Title: Coexistence HBsAg/HBcAC, Clinical Characterístics & Outcomes
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Consorci Sanitari de Terrassa (Other); Hospital Universitario La Fe (Other); Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Mireia Miquel-Planas, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2022/5032
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Not apply: None. Just registration epidemiology dates

SUMMARY:
HBV infection is a dynamic process with complex interactions between virus replication and the host's immune response. The appearance of anti-HBs after HBV infection generally indicates recovery and immunity to HBV1 infection. However, there are several published studies that describe the coexistence of the marker of chronic infection (HBsAg +) and the marker of functional cure (HBsAc +). There are contradictory studies on whether the coexistence of HBsAg/HBsAc implies a different clinical course.

ELIGIBILITY:
Inclusion Criteria:

* all those patients who have been seen in outpatient hepatology consultations and who present positive HBsAg and HBsAc serology simultaneously.

Exclusion Criteria:

* Hepatitis C or HIV Co-infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All those patients included all patients visited asoutpatient hepatology consultations of the respective centers in the last 10 years (between 01/01/2010 and 12/31/2020) and who present positive HBsAg and HBsAc serology simultaneously.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence concomitant HBsAg and HBsAc markers | 10 years
  To describe the prevalence of concomitant HBsAg and HBsAc markers in our area

SECONDARY OUTCOMES:
differences between immunocompetent patients with respect to immunocompromised ones. | 10 years
  To compare if there are differences in the prevalence or clinical outcome according if the patient has any degree of immunosupresion or not.

CONTACTS AND LOCATIONS:
Locations (1):
- H. Consorci Sanitari Parc Tauli, Sabadell, Barcelona, Spain